CLINICAL TRIAL: NCT05021042
Title: Identification of Predictive Biomarkers of Mastitis in Lactating Mothers Using a Metabolomic Approach
Brief Title: Identification of Biomarkers of Mastitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LactApp Women's Health (Industry)
Responsible Party: Principal Investigator, Paola Quifer Rada, Clinical Data Researcher, LactApp Women's Health
Other Study IDs: LactApp001
Record Dates: First submitted 2021-08-11; First posted 2021-08-25 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Breast Feeding; Mastitis; Mastitis Acute Female
Keywords: breastfeeding; breast milk; mastitis; acute mastitis; subacute mastitis; biomarkers
MeSH Terms: conditions — Breast Feeding; Mastitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute mastitis (MA): Lactating women with confirmed acute mastitis
- Subacute mastitis (SAM): Lactating women with confirmed subacute mastitis
- Control (CT): Lactating women with the absence of acute or subacute mastitis symptomatology.

SUMMARY:
Breastfeeding is the optimal feeding for infants. WHO currently promotes breastfeeding and recommends it to be exclusive until the baby is 6 months old. Breastfeeding has a positive impact on both the mother's and the infant's health and is directly associated with the decrease in diseases such as cancer, diabetes, cardiovascular disease, and inflammatory and infectious diseases. Currently, in Spain, only 39% of infants at 6 months are breastfed. The factors that influence the abandonment of breastfeeding are returning to work, the sensation of hypogalactia, problems to breastfeed, and breast complications, like mastitis, being the pain its main cause. Recent studies have associated pain while breastfeeding with mammary gland inflammation (mastitis) caused by dysbiosis.

In order to increase breastfeeding rates, it is necessary to find factors related to the progression of mastitis in breastfeeding women. In this context, the discovery of predictive biomarkers based on metabolic markers is key to act before or at the beginning of the progression of mastitis and thus reduce the rates of abandonment of breastfeeding due to pain.

The present project aims to identify and validate metabolic biomarkers capable of predicting mastitis. For this purpose, a prospective observational case-control hypothesis-free study will be carried out in order to identify and validate biomarkers of mastitis in breastfeeding women. The study will be performed in two phases: the discovery of the possible biomarkers and the validation of the biomarkers.

Breast milk will be collected at the beginning of the study and when women present symptoms compatible with mastitis. The presence or not of mastitis will be confirmed with a milk culture. Milk samples will be analyzed using non-targeted metabolomics approach. Using multivariate statistical models, the potential metabolites capable of discriminating the presence of mastitis in maternal milk will be identified. Later, these potential markers will be validated in independent samples.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding women with healthy full-term, singleton infants older than 1 months weeks and younger than 6 months.
* Provide written informed consent

Exclusion Criteria:

* Immunocompromised suppressed women (i.e. HIV, following treatment with immunosuppressants or chemotherapy).
* Currently being treated for cancer
* Current infection being treated with antibiotics.
* Women who carry out a complete deferred breastfeeding.
* Women with babies presenting any syndrome, cleft lip or facial malformations.
* Currently tandem breastfeeding.
* Women who have had a premature delivery

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Lactating women will be included in the study. Women with the presence of acute mastitis, subacute mastitis, and with absence of symptomatology compatible with mastitis will be recruited as control samples.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Breast milk metabolites | 6 months
  Breast milk Metabolite will be identified by NMR metabolomic analysis. Analytes will be quantified in mg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- LactApp Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://lactapp.com/